CLINICAL TRIAL: NCT04385953
Title: Evaluation of the Clinical Performance of the Quantra System With the QStat Cartridge in Trauma and Obstetric Hemorrhage
Brief Title: QStat in Trauma and Obstetric Hemorrhage
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-030
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Blood Loss Massive; Trauma; Post Partum Hemorrhage
Keywords: Viscoelastic testing; Coagulation; Quantra; Hemostasis
MeSH Terms: conditions — Wounds and Injuries; Postpartum Hemorrhage; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Trauma patients: Subject experiencing major trauma
  Interventions: Diagnostic Test: Quantra System
- Obstetric patients: Obstetric patient with postpartum hemorrhage
  Interventions: Diagnostic Test: Quantra System

INTERVENTIONS:
Diagnostic Test: Quantra System — Diagnostic device to monitor coagulation properties of a whole blood sample at the point-of-care
  Other Names: Quantra QStat Cartridge

SUMMARY:
This study will evaluate the performance of the Quantra System comprised of the Quantra Hemostasis Analyzer with the QStat Cartridge in trauma patients and obstetric patients with postpartum hemorrhage.

DETAILED DESCRIPTION:
The Quantra System is a fully integrated and automated in vitro diagnostic device which uses SEER Sonorheometry, an ultrasound-based technology, to characterize the viscoelastic properties of a whole blood sample during coagulation. The QStat Cartridge was developed to monitor hemostasis in patients that may experience a range of coagulopathies of various etiologies including fibrinolytic defects. This includes the trauma, obstetric hemorrhage and liver transplant populations. The cartridge consists of four independent channels each containing different sets of reagents, which provide four measurements performed in parallel yielding five parameters that depict the functional status of a patient's coagulation system.

This prospective, observational pilot study will evaluate the performance of the Quantra System with the QStat Cartridge as compared to comparable measures using conventional viscoelastic testing methods.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age
* Subject is a trauma patient experiencing major trauma (preferably requiring the highest level of team activation) with active bleeding or deemed at high risk of significant bleeding according to mechanism of injury.and is a candidate for a ROTEM test to be performed to access coagulopathy.

OR

-Subject is an obstetric patient experiencing post-partum hemorrhage based on one of the following conditions: estimated blood loss during delivery >1000 mL; placental abruption with hemorrhage of any quantity; clinically suspected DIC; pregnancy resulted in fetal demise with hemorrhage of any quantity; or is under consideration for administration of tranexamic acid for treatment of hemorrhage.

Exclusion Criteria:

* Subject is younger than 18 years of age
* Subject presents for a procedure intended to abort a pregnancy for reasons other than medical necessity
* Subject is known to have received antifibrinolytic therapy immediately prior to presentation to trauma unit
* Subject is currently enrolled in a distinct study that might confound the results of the proposed study
* Subject is affected by a condition that, in the opinion of the clinical team, may pose additional risks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential study participants will be adult (>18 years) trauma patients or obstetric patients with postpartum hemorrhage where visicoelastic testing is performed as standard of care to assess coagulopathy.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the Quantra results to corresponding ROTEM Delta results | Upon arrival to emergency department
  Coagulation function assessed by Quantra and ROTEM delta
Comparison of the Quantra results to corresponding ROTEM Delta results | At the time of hemorrhage for obstetric patients
  Coagulation function assessed by Quantra and ROTEM delta

CONTACTS AND LOCATIONS:
Locations (1):
- Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No